CLINICAL TRIAL: NCT00583648
Title: A Randomized Controlled Trial Showing the Effect of Patient Lenght of Stay in the Emergency Department Through Utilizing a Urinalysis Nursing Protocol.
Brief Title: Does Implementing a Urinanylsis Protocol Based on Symptoms Decrease Length of Stay in the Emergency Department?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, David Schriger, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: UCLA-urineprotocol; UCLA-12345
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Urinary Tract Infections
Keywords: urinary tract infections; urine; urinalysis; urine protocols; urinalysis protocols; nursing protocols; Emergency Department
MeSH Terms: conditions — Urinary Tract Infections; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Recieves urinalysis by nurse per set protocol based off of inclusion criteria
  Interventions: Other: Urinanlysis
- 2 (No Intervention): ordering of test will be up to the treating physician

INTERVENTIONS:
Other: Urinanlysis — sending a Urine sample to the laboratory for processing
  Other Names: UA
  Arms: 1

SUMMARY:
The implementation of nursing urinanlysis protocols based off of symptoms of urinary infections will significantly decrease the length of a patient's stay in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* patients between 16 and 65 years of age complaining of any of the following: dysuria, hematuria, urinary frequency, urinary urgency

Exclusion Criteria:

* any person less than 16 or greater than 65 years of age, history of kidney disease or transplant, foley catherization within the last 30 days, on immuno-suppresent and/or receiving chemotherapy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Length of Stay in the Emergency Department | 1 hour

SECONDARY OUTCOMES:
Physician decision making on ordering urinalysis based off of chief complaints | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Seefeld, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles Medical Center, Los Angeles, California, United States